CLINICAL TRIAL: NCT05348096
Title: Efficacy and Safety of the Combination of Low-dose Ibrutinib and Itraconazole in Moderate to Severe Chronic Graft Versus Host Disease: a Phase 2 Trial
Brief Title: Efficacy and Safety of Low-dose Ibrutinib and Itraconazole in Chronic Graft Versus Host Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Cesar Homero Gutierrez-Aguirre, Clinical Professor, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI22-00027
Record Dates: First submitted 2022-04-13; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Chronic Graft-versus-host-disease
Keywords: ibrutinib; low-dose; azole; itraconazole; refractory
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — ibrutinib

STUDY DESIGN:
Intervention Model Description: Patients will receive oral ibrutinib (140mg QD) combined with a CYP3A4 inhibitor (oral itraconazole, 100mg BID) for six months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-dose ibrutinib (Experimental): Patients will receive ibrutinib 140mg/day PO in combination with oral itraconazole (100mg/day) continuously for six months.
  Interventions: Drug: Low-dose ibrutinib

INTERVENTIONS:
Drug: Low-dose ibrutinib — Daily ibrutinib (140mg QD) and itraconazole (100mg BID) for six months.
  Other Names: INN-ibrutinib

SUMMARY:
Chronic graft-versus-host disease (cGVHD) affects 30 to 70% of Allogeneic Hematopoietic Cell Transplantation, decreases the quality of life, and increases mortality. First-line treatments for cGVHD are steroids, however, up to 50% of patients do not respond to treatment. There is no well-defined second-line treatment for cGVHD, but ibrutinib, a Bruton tyrosine kinase inhibitor, has been successfully used in phase 2 clinical trials for moderate to severe steroid-refractory cGVHD and has been shown to be safe, showing rates of response of 69% at a median follow-up of 26 months. Therefore, ibrutinib was approved by the FDA for the treatment of steroid-refractory cGVHD. Also, it is known that ibrutinib is metabolized by cytochrome isoenzyme 3A4 and that itraconazole is a potent inhibitor of this hepatic isoenzyme. Therefore, the investigators hypothesized that in subjects with newly diagnosed cGVHD and in patients with steroid-refractory cGVHD, low-dose ibrutinib in combination with itraconazole might be effective and safe.

DETAILED DESCRIPTION:
In this phase 2 clinical trial, patients with newly diagnosed cGVHD and refractory cGVHD will receive low-dose ibrutinib (140mg/day) combined with a cytochrome 3A4 inhibitor (itraconazole, 100mg BID) for six months. The follow-up consists of weekly visits for the first months and then monthly for six months. The investigators will address clinical and biochemical parameters in each visit and grade severity using the NIH (2014) scale. Also, patients will answer the modified Lee symptom scale, and grade response to treatment using the National Institutes of Health (NIH) Consensus Panel Chronic GVHD Activity Assessment (2014). The investigators will grade adverse events with the Common Terminology Criteria for Adverse Events [v5.0]. The investigators will report proportion and time to any response, complete response, partial response, stable disease, and progression. Also, the investigators will report the proportion of patients that interrupted steroids for at least one month, the proportion of patients that interrupted every immunosuppressive therapy for at least one month, and the proportion of patients that interrupted ibrutinib specifying the cause of the interruption.

ELIGIBILITY:
Inclusion Criteria:

* Age (>18 years)
* Any type of peripheral blood stem cell transplant (matched-related, match non-related, and haplo)
* Any conditioning regimen
* Newly diagnosed moderate to severe chronic graft versus host disease
* Steroid refractory moderate to severe chronic graft versus host disease defined as progression with prednisone 1mg/kg/day, or stable disease after four to six weeks of prednisone >0.5 mg/kg/day, or disease progression when reducing prednisone below <0.5 mg/kg/día.

  5. Eastern Cooperative Oncology Group (ECOG) <= 2

Exclusion Criteria:

* Disease relapse (excluding positive minimal residual disease)
* Secondary malignancies
* Disease progression
* Use of B lymphocyte cytotoxics in the last month (i.e., rituximab, bortezomib)
* Advance stages of heart failure (NYHA III o IV)
* Ventricular arrhythmias
* Uncontrolled hypertension
* Ischemic heart diseases such as unstable angina or stable angina in the last six months
* Hepatitis B or C
* Hypersensitivity to ibrutinib
* Active bleeding
* Uncontrolled acute infection
* Hepatopathy Child-Pugh C
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Treatment safety | Up to six months of enrollment
  Treatment safety will be addressed by obtaining the proportion of patients with grade >=3 adverse events as defined by the Common Terminology Criteria for Adverse Events [v5.0]. If the proportion of >=3 adverse events is less than 20% then the treatment will be defined as safe.
Overall response rate | Up to six months of enrollment
  The proportion of patients with partial and/or complete response at six months of follow-up.

SECONDARY OUTCOMES:
Overall treatment-free survival | Up to six months post enrollment
  The proportion of patients with any other treatment rather than ibrutinib at six months of follow-up.
Steroid-free cumulative incidence | Up to six months post enrollment
  The number of patients using 0mg of prednisone for at least one month divided by the total number of patients at the time interval of the study.
Low-dose steroid cumulative incidence | Up to six months post enrollment
  The number of patients using less than 0.15 mg/kg/day of prednisone 0 for at least one month divided by the total number of patients at the time interval of the study.
Immunosuppressive-free cumulative incidence | Up to six months post enrollment
  The number of patients without any immunosuppressor divided by the total number of patients at the time interval of the study.
Overall survival | Up to six months post enrollment
  Overall survival is defined as the length of time from the start of ibrutinib to the time of death.
Time to any response | From date of inclusion until the date of first documented response (partial or complete), assessed up to six months.
  Time length from the first day of ibrutinib to any response (partial response or complete response)
Time to progression | From date of inclusion until the date of first documented progression, assessed up to 6 months.
  Time length from the first day of ibrutinib to progression.
Complete response rate | Up to six months post enrollment
  The complete response rate was defined as the proportion of patients that achieve complete responses within the study's time frame.
Partial response rate | Up to six months post enrollment
  The partial response rate was defined as the proportion of patients that achieve partial responses within the study's time frame.
Progression rate | Up to six months post enrollment
  The progression rate was defined as the proportion of patients that progresses within the study's time frame.
Any adverse events rate | Up to six months post enrollment
  The any adverse event rate was defined as the proportion of patients with any grade adverse events within the study's time frame.
Proportion of therapy interruption | Up to six months post enrollment
  The proportion of patients that need ibrutinib interruption because of unacceptable toxicity (grade >=3).

CONTACTS AND LOCATIONS:
Overall Officials: Fernando De la Garza Salazar, Principal Investigator — Hospital Universitario Dr. José Eleuterio González
Locations (1):
- Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolff D, Fatobene G, Rocha V, Kroger N, Flowers ME. Steroid-refractory chronic graft-versus-host disease: treatment options and patient management. Bone Marrow Transplant. 2021 Sep;56(9):2079-2087. doi: 10.1038/s41409-021-01389-5. Epub 2021 Jul 3. PMID 34218265
- [Result] Waller EK, Miklos D, Cutler C, Arora M, Jagasia MH, Pusic I, Flowers MED, Logan AC, Nakamura R, Chang S, Clow F, Lal ID, Styles L, Jaglowski S. Ibrutinib for Chronic Graft-versus-Host Disease After Failure of Prior Therapy: 1-Year Update of a Phase 1b/2 Study. Biol Blood Marrow Transplant. 2019 Oct;25(10):2002-2007. doi: 10.1016/j.bbmt.2019.06.023. Epub 2019 Jun 28. PMID 31260802
- [Result] Tapaninen T, Olkkola AM, Tornio A, Neuvonen M, Elonen E, Neuvonen PJ, Niemi M, Backman JT. Itraconazole Increases Ibrutinib Exposure 10-Fold and Reduces Interindividual Variation-A Potentially Beneficial Drug-Drug Interaction. Clin Transl Sci. 2020 Mar;13(2):345-351. doi: 10.1111/cts.12716. Epub 2019 Nov 29. PMID 31664782